CLINICAL TRIAL: NCT06005909
Title: Investigation of the Effects of Exercises With Mechanical Hippotherapy Device and Cawthorne-Cooksey Exercises on Balance, Dizziness, Fatigue and Quality of Life in Patients With Multiple Sclerosis.
Brief Title: Current Exercise Approaches in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar62
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
Keywords: Dizziness; Cawthorne-Cooksey; Hippotherapy simulator; Balance; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Dizziness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cawthorne-Cooksey (Experimental): These exercises, which are designed to reduce vertigo, stabilize the gaze and improve balance by stimulating or operating the vestibular system during daily activities, consist of a series of eye, head, trunk and balance movements that provoke vestibular symptoms and whose difficulty increases. The degree of difficulty of the exercises was increased with the improvement of the patient. Head and trunk movements while sitting, standing and walking were added to the exercises that initially started with simple eye-head movements in bed.
  Interventions: Other: Cawthorne-Cooksey Exercises
- Mechanical Hippotherapy (Experimental): Before being taken to the device, the patients were informed about the working principle of the device, the exercises to be performed on the device, and that the exercise would be terminated in case of a possible health problem. After being placed on the device, the patient was given time until the initial balance was achieved. When the patient felt ready, a 15-minute hippotherapy session was applied at the 5th level of the 20-stage speed level by the physiotherapist.
  Interventions: Other: Mechanical Hippotherapy Exercises

INTERVENTIONS:
Other: Cawthorne-Cooksey Exercises — A- Head and Eye Movements While Lying and Sitting:
  1. While keeping your head still, look up and then down again.
  2. Look from side to side while keeping your head still.
  3. Extend your hand at arm's length, draw your fingers towards your nose while focusing your eyes on your fingers.
  4. With eyes open, slowly turn your head from side to side.
  5. Turn your head from side to side quickly.
  6. With eyes open, slowly move your head up and down.
  7. Move your head up and down quickly.
  8. Repeat items 4,5,6 and 7 with your eyes closed.
  B-Head and Body Movements While Sitting:
  1. Place an object on the floor in front of your feet, reach out to pick it up, then upright return to your position. Looking down while picking up the item, then Remind you to look up when trying to fix it.
  2. Lean forward and move the object forward and back under your knees. C- Standing Exercises
  1-Get from a sitting position to a standing position and sit down again. 2-Repeat this with your eyes closed.
  Arms: Cawthorne-Cooksey
Other: Mechanical Hippotherapy Exercises — From the patient on the mechanical hippotherapy device;
  * Maintaining trunk balance while raising both hands above head,
  * Maintaining trunk balance while opening the arms next to the trunk,
  * Maintaining trunk balance while extending the arms back and forth with successive movements,
  * Maintaining trunk balance with hands clasped behind the waist,
  * The arms are open to both sides, while transferring the weight ball from one hand to the other, it is requested to maintain the body balance.
  Arms: Mechanical Hippotherapy

SUMMARY:
This study was conducted to examine the effects of exercises performed with mechanical hippotherapy device and Cawthorne-Cooksey exercises on balance, dizziness, fatigue and quality of life in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
The research is a quantitative study, and it is in the form of randomized controlled type research, one of the experimental research types. In order to provide a homogeneous distribution, the patients were divided into two different exercise groups using the double-blind method from the minimization method.

The sample of the study consisted of definitively diagnosed multiple sclerosis (MS) patients who volunteered to participate in the study. Patients who voluntarily agreed to participate in the study; While they were informed about the aims of the study, the duration of the study, the evaluation methods and the applications to be made, the informed consent form was signed by these patients and their consent was obtained. The study sample was divided into two groups by randomization method. The first group was given 35 minutes of traditional physical therapy program and 15 minutes of exercises with a mechanical hippotherapy device, while the second group was given 15 minutes of Cawthorne-Cooksey exercises in addition to the 35-minute traditional physical therapy program. Both exercise groups were given a 50-minute physical therapy program. Patients diagnosed with Multiple Sclerosis in the study; It was classified according to the Expanded Disability Status Scale Score. Tinetti Balance Rating Scale was used to assess balance. The Dizziness Disability Inventory was used to assess dizziness, the Fatigue Severity Scale and the Fatigue Impact Scale to assess fatigue, and the Ferrans & Powers Quality of Life Index MS Adaptation to assess quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being cooperative and oriented,
* Being 25 - 64 years
* Having a definite diagnosis of MS,
* Being able to sit dependent/independently and stand supported/unsupported,
* Not having an attack in the last 1 month or not currently in the attack period,
* Volunteering to participate in the study.

Exclusion Criteria:

* Having another neurological disease or musculoskeletal system problems in addition to the diagnosis of MS,
* Being on cortisone treatment in the last 1 month or still ongoing,
* Having a mental, cardiovascular, pulmonary or orthopedic disease that will prevent exercise.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Fatigue severity scale | 10 weeks
  The lowest score that can be obtained from the scale is 9, and the highest score is 63. The fatigue severity scale is the average value of nine sections. A high score indicates increased fatigue severity. The scale, including the day it was filled, questions the state of fatigue in the last 1 month.
Fatigue Impact Scale | 10 weeks
  The scale consists of 40 questions. The first 10 items evaluate the cognitive state, the second 10 items evaluate the physical state, and the third 20 items evaluate the psychological state. Participants gave each question a score between 0 (no problem) and 4 (maximum problem). The highest score is 160. High scores indicate fatigue. The scales question the state of fatigue in the last 1 month, including the day it was filled in. The fatigue impact scale was found to be the most ideal scale to evaluate the effect of fatigue on daily life in MS.
Tinetti balance rating scale | 10 weeks
  The scale includes gait (AS) and balance (EP) subgroups. Evaluation is made with specific scoring criteria for each activity. The total score is a maximum of 28, including the walking subgroup score and the balance subgroup score. The scores obtained by the participants were recorded separately for walking and balance, and the total score was also written. Scores of 18 and below are associated with high, scores between 19 and 23 are associated with moderate, and scores of 24 and above are associated with a low risk of falling.
Dizziness disability inventory | 10 weeks
  The participants were asked to score this inventory, which consists of 25 items, according to the frequency and severity of the vertigo complaint and the degree of impact it creates in daily life. Sub-inventories are intended to determine the physical, sensory and functional effects of vestibular system diseases. In the scoring of the sub-units of the inventory, 28 points determine physical disability, 36 points functional and sensory disability. The scores obtained were recorded as physical disability, emotional disability and functional disability data. The final result consists of the sum of all of them. High scores are interpreted as the patient's vertigo complaint preventing his further life.
Ferrans&Powers quality of life index | 10 weeks
  This index has 5 subcategories. These; total quality of life score, health and functionality subcategory score, social and economic subcategory score, psychological/belief subcategory score and family subcategory score. The test has two parts, satisfaction and importance, and each part has the same number of questions, question content is the same. The participants were asked to fill in the questionnaire and the physiotherapist calculated the values in accordance with the scoring instructions. The score of these collected values was divided by the number of marked questions. The final score was obtained by adding 15 to the obtained values. The final score is between 0-30.
Extended disability status scale | 10 weeks
  In the Disability Status Scale, the patient is evaluated over a total of 10 points. While zero indicates normal health status, 10 indicates death due to an uncommon Multiple Sclerosis. In this scale, which consists of twenty steps, 0 indicates normal neurological finding; 10 means death due to MS. Scores on the Extended disability status scale increase to correspond with worsening in MS. The first score after 0 is 1, and then clinical worsening is expressed in 0.5-point intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Alesta KABUK, Study Chair — Uskudar University
Locations (1):
- Baskent University Istanbul Hospital, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coban O, Mutluay F. The effects of mechanical hippotherapy riding on postural control, balance, and quality of life (QoL) in patients with stroke. Disabil Rehabil. 2024 Jun;46(11):2338-2347. doi: 10.1080/09638288.2023.2221458. Epub 2023 Jun 11. PMID 37303153
- [Background] Tacalan E, Inal HS, Senturk MN, Mengi E, Alemdaroglu-Gurbuz I. Effectiveness of the Epley maneuver versus Cawthorne-Cooksey vestibular exercises in the treatment of posterior semicircular canal benign paroxysmal positional vertigo (BPPV): A randomized controlled trial. J Bodyw Mov Ther. 2021 Oct;28:397-405. doi: 10.1016/j.jbmt.2021.07.030. Epub 2021 Aug 8. PMID 34776169
- [Background] Afrasiabifar A, Karami F, Najafi Doulatabad S. Comparing the effect of Cawthorne-Cooksey and Frenkel exercises on balance in patients with multiple sclerosis: a randomized controlled trial. Clin Rehabil. 2018 Jan;32(1):57-65. doi: 10.1177/0269215517714592. Epub 2017 Jun 19. PMID 28629268